CLINICAL TRIAL: NCT05141513
Title: A Safety Study of Intraoperative Radiation Therapy Following Stereotactic Body Radiation Therapy and Multi-agent Chemotherapy in the Treatment of Localized Pancreatic Adenocarcinoma
Brief Title: Intraoperative Radiation Therapy After Stereotactic Body Radiation Therapy and Chemotherapy in Treatment of Pancreatic Adenocarcinoma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: J21105; IRB00294801 (Other: Johns Hopkins Medicine)
Record Dates: First submitted 2021-11-23; First posted 2021-12-02 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Intervention Model Description: This is a prospective, single institution, single arm pilot study to evaluate the safety and feasibility of implementing IORT in patients with non-metastatic Pancreatic adenocarcinoma (PDAC) who have been treated with neoadjuvant chemotherapy and SBRT and who are undergoing surgical resection.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Intra Operative Radiation Therapy (IORT) Group (Other): The IORT group is the single arm of this study. Enrolled patients who undergo standard of care treatment will also receive a study treatment of High Dose Rate (HDR) Intra Operative Radiation Therapy.
  Interventions: Radiation: High Dose Rate Brachytherapy (HDR) Intraoperative Radiation Therapy (IORT)

INTERVENTIONS:
Radiation: High Dose Rate Brachytherapy (HDR) Intraoperative Radiation Therapy (IORT) — After the patient receives standard of care treatment, they will receive a single dose of radiation (15 Gy) at the time the tumor is surgically removed. Surgeons will then place clips along the blood vessels around the surgical area. These clips will be used to confirm (after surgery) that the expected dose of radiation was received during surgery.

SUMMARY:
This study is designed to investigate the safety of intraoperative radiation therapy (IORT) in patients with localized pancreatic cancer undergoing surgical resection after neoadjuvant chemotherapy and stereotactic body radiation therapy (SBRT).

DETAILED DESCRIPTION:
Standard of care treatment for patients with non-metastatic pancreatic adenocarcinoma (PDAC) includes chemotherapy and Stereotactic Body Radiation Treatment (SBRT) followed by surgical resection of the tumor with or without Intra-Operative Radiation Therapy (IORT).

There is some evidence from other research studies suggesting that adding radiation treatment during the surgical resection may improve local control of the cancer. The use of IORT plus surgical resection can be used to treat pancreatic cancer and is done on a case by case basis at Johns Hopkins.

The department of Radiation Oncology has developed a program using a High Dose Rate-IORT (HDR-IORT). The HDR-IORT makes it possible to deliver concentrated radiation dose at the surface of the tumor.

Our team has shown in previous studies that the majority of cancer cells that remain after treatment are located around the area of the pancreas called the "Triangle Volume" (TV). This region contains blood vessels, lymphatic vessels, and nerves, and is at high risk of containing cancer cells. This region is difficult to treat with SBRT alone because of being close to normal, healthy organs. Therefore, this study involves using IORT to treat the TV to a therapeutic radiation dose.

The part of the treatment that is considered research is:

* Giving one dose of 15 Gy during the surgery using IORT to deliver radiation, and
* Targeting the larger area around the pancreas called the TV

The goal of this study is to determine safety of this added treatment which will be assessed at 3 months after the surgery is completed.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years old
2. Resectable/BRPC/LAPC as defined by NCCN guidelines (Figure 1) as follows confirmed via CT, EUS, or other imaging modalities.
3. ECOG performance status 0-2
4. Subject or authorized representative, has been informed of the nature of the study and has provided written informed consent, approved by the appropriate Institutional Review Board (IRB) of the respective clinical site.
5. Candidate for SBRT at JHU
6. Upfront treatment with multi-agent chemotherapy
7. Candidate for surgical exploration at JHU

Exclusion Criteria:

1. Previous thoracic/abdominal radiation therapy
2. Unable to receive SBRT at JHU
3. Duodenal invasion detected on imaging which would exclude candidacy for SBRT
4. Tumor located in pancreatic body or tail
5. Unable to undergo Whipple procedure
6. Evidence of disease not localized to the pancreas
7. Any arterial reconstruction during surgery
8. Currently enrolled in another investigational drug or device trial that clinically interferes with this study
9. Unable to comply with study requirements or follow-up schedule
10. Women of child bearing potential or sexually active fertile men with partners who are women of child bearing potential who are unwilling or unable to use an acceptable method to avoid pregnancy for the entire study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2022-05-06 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
Acute post-operative toxicity of targeted IORT | 3 months
  To evaluate acute post-operative toxicity of IORT targeted to the TV in patients with non-metastatic PDAC undergoing surgical resection after neoadjuvant multi-agent chemotherapy and SBRT.

SECONDARY OUTCOMES:
Late post-operative toxicity of targeted IORT | 6 months
  To evaluate late toxicity of IORT targeted to the TV in patients with non-metastatic PDAC undergoing surgical resection after neoadjuvant multi-agent chemotherapy and SBRT.
  To evaluate late toxicity (>90 days) of IORT targeted to the TV in patients with non-metastatic PDAC undergoing surgical resection after neoadjuvant multi-agent chemotherapy and SBRT.
Late post-operative toxicity of targeted IORT | 12 months
  To evaluate late toxicity of IORT targeted to the TV in patients with non-metastatic PDAC undergoing surgical resection after neoadjuvant multi-agent chemotherapy and SBRT.
  To evaluate late toxicity (>90 days) of IORT targeted to the TV in patients with non-metastatic PDAC undergoing surgical resection after neoadjuvant multi-agent chemotherapy and SBRT.
Late post-operative toxicity of targeted IORT | 24 months
  To evaluate late toxicity of IORT targeted to the TV in patients with non-metastatic PDAC undergoing surgical resection after neoadjuvant multi-agent chemotherapy and SBRT.
  To evaluate late toxicity (>90 days) of IORT targeted to the TV in patients with non-metastatic PDAC undergoing surgical resection after neoadjuvant multi-agent chemotherapy and SBRT.
Late post-operative toxicity of targeted IORT | 36 months
  To evaluate late toxicity of IORT targeted to the TV in patients with non-metastatic PDAC undergoing surgical resection after neoadjuvant multi-agent chemotherapy and SBRT.
  To evaluate late toxicity (>90 days) of IORT targeted to the TV in patients with non-metastatic PDAC undergoing surgical resection after neoadjuvant multi-agent chemotherapy and SBRT.
Median local-progression free survival (LPFS) from IORT | 6 months
  To determine the median local-progression free survival (LPFS) from time of IORT.
Median local-progression free survival (LPFS) from IORT | 12 months
  To determine the median local-progression free survival (LPFS) from time of IORT.
Median local-progression free survival (LPFS) from IORT | 24 months
  To determine the median local-progression free survival (LPFS) from time of IORT.
Median local-progression free survival (LPFS) from IORT | 36 months
  To determine the median local-progression free survival (LPFS) from time of IORT.
Median overall survival (OS) from IORT | 6 months
  To determine the median overall survival (OS) from time of IORT.
Median overall survival (OS) from IORT | 12 months
  To determine the median overall survival (OS) from time of IORT.
Median overall survival (OS) from IORT | 24 months
  To determine the median overall survival (OS) from time of IORT.
Median overall survival (OS) from IORT | 36 months
  To determine the median overall survival (OS) from time of IORT.
Median progression free survival (PFS) from IORT | 6 months
  To determine the median progression free survival (PFS) from time of IORT
Median progression free survival (PFS) from IORT | 12 months
  To determine the median progression free survival (PFS) from time of IORT
Median progression free survival (PFS) from IORT | 24 months
  To determine the median progression free survival (PFS) from time of IORT
Median progression free survival (PFS) from IORT | 36 months
  To determine the median progression free survival (PFS) from time of IORT

CONTACTS AND LOCATIONS:
Overall Officials: Amol Narang, MD, Principal Investigator — JHU, School of Medicine, SKCCC
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Reddy AV, Hill CS, Zheng L, He J, Narang AK. A safety study of intraoperative radiation therapy following stereotactic body radiation therapy and multi-agent chemotherapy in the treatment of localized pancreatic adenocarcinoma: study protocol of a phase I trial. Radiat Oncol. 2022 Oct 28;17(1):173. doi: 10.1186/s13014-022-02145-9. PMID 36307845